CLINICAL TRIAL: NCT01960192
Title: The Prospective Study of FVD Program and HD-MTX-Ara-C Program Contrast in the Treatment of PCNSL Lymphoma.
Brief Title: Treatment of Primary CNS Lymphoma
Acronym: FVD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Collaborators: Zhengzhou University (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2011-6
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Primary CNS Lymphoma (PCNSL)
Keywords: primary CNS lymphoma;chemotherapy;; RR;PFS;OS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FVD regimen (Experimental): FVD regimen(fotemustine, teniposide and dexamethasone),fotemustine 100mg/m2 d1 ivgtt,teniposide 60mg/m2 d2-4 ivgtt,dexamethasone 40mg d1-5 ivgtt.Continued use to the end of chemotherapy .Every 21 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles.
  Interventions: Drug: FVD regimen
- HD-MTX-Ara-C regimen (Experimental): high-does metrotrexate 3.5g/m2 d1 ivgtt 6h,cytarabine 1g/m2 bid d2-3.Continued use to the end of chemotherapy .Every 21 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles.
  Interventions: Drug: HD-MTX-Ara-C regimen

INTERVENTIONS:
Drug: HD-MTX-Ara-C regimen — high-does metrotrexate 3.5g/m2 d1 ivgtt 6h,cytarabine 1g/m2 bid d2-3.Continued use to the end of chemotherapy .Every 21 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles
  Arms: HD-MTX-Ara-C regimen
Drug: FVD regimen — FVD regimen(fotemustine, teniposide and dexamethasone),fotemustine 100mg/m2 d1 ivgtt,teniposide 60mg/m2 d2-4 ivgtt,dexamethasone 40mg d1-5 ivgtt.Continued use to the end of chemotherapy .Every 21 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles
  Arms: FVD regimen

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of FVD regiment (fotemustine, teniposide and dexamethasone ) for patients with primary CNS lymphoma.

DETAILED DESCRIPTION:
Primary CNS lymphoma (PCNSL) is a rare B-cell variant of non-Hodgkin lymphoma that is confined to the brain, leptomeninges, spinal cord, and eyes. The optimum treatment for patients with PCNSL remains challenging and at present there is no universally accepted therapeutic approach for patients with newly diagnosed disease. The purpose of this study is to evaluate the efficacy and safety of FVD regiment(fotemustine, teniposide and dexamethasone)contrast with HD-MTX-Ara-C program for patients with primary CNS lymphoma.

ELIGIBILITY:
Inclusion Criteria:Age range 14-60 years old; ECOG performance status 0-2; Estimated survival time > 3 months Histological confirmed PCNSL None of chemotherapy or radiotherapy has been previously used None of chemotherapy contraindication: hemoglobin ≥ 90 g/dl, neutrophil ≥ 1.5×109/L, platelet ≥ 100×109/L, ALT and AST ≤ 2×ULN, serum bilirubin ≤ 1.5×ULN, serum creatine ≤ 1.5×upper limitation of normal (ULN), Serum Albumin ≥ 30g/L, serum plasminogen is normal (Inclusion Criteria of 1,3,6 groups ) At least one measurable lesion None of other serious diseases, cardiopulmonary function is normal Pregnancy test of women at reproductive age must be negative Patients could be followed up None of other relative treatments including the traditional Chinese medicine, immunotherapy,biotherapy except anti-bone metastasis therapy and other symptomatic treatments.

volunteers who signed informed consent. -

Exclusion Criteria:Disagreement on blood sample collection Patients allergic of any of drug in this regimen or with metabolic disorder Pregnant or lactating women Serious medical illness likely to interfere with participation Serious infection Primitive or secondary tumors of central nervous system Chemotherapy or radiotherapy contraindication The evidence of peripheral nervous disorder or dysphrenia patients participating in other clinical trials patients taking other antitumor drugs patients estimated to be unsuitable by investigato

-

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to end of follow-up-phase (approximately 24 months)

SECONDARY OUTCOMES:
response rate | every 6 weeks,up to completion of treatment(approximately 18 weeks )
overall survival | up to the date of death (approximately 5 years)
median survival time | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Pro,Dr, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China